CLINICAL TRIAL: NCT03202355
Title: The Effect of OrthoPulse Photobiomodulation on the Rate of Tooth Movement During Alignment With Fixed Appliances
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated due to clinical staffing changes and enrolment
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BX11
Record Dates: First submitted 2017-06-19; First posted 2017-06-28 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Malocclusion
Keywords: Alignment phase; Photobiomodulation; Orthodontic treatment; Malocclusion; OrthoPulse™
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel, open-label, non-randomized, controlled, private practice study designed to evaluate the intended purposes of the investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Control) (Experimental): Subjects assigned to this group receive fixed appliance orthodontic treatment only
  Interventions: Device: Fixed Appliance Orthodontic Treatment
- Group 2 (OP1) (Experimental): Subjects assigned to this group receive fixed appliance orthodontic treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Interventions: Device: Fixed Appliance Orthodontic Treatment; Device: OrthoPulse™

INTERVENTIONS:
Device: Fixed Appliance Orthodontic Treatment — Patients receive fixed appliance orthodontic treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
Device: OrthoPulse™ — Patients carry out daily OrthoPulse™ treatments at home.
  Arms: Group 2 (OP1)

SUMMARY:
The aim of this study is to determine efficacy of OrthoPulse photobiomodulation on the rate of tooth movement during alignment for Subjects receiving fixed appliance orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of permanent dentition
* Eligible and scheduled for full-mouth, fixed-appliance orthodontic treatment
* Moderate to severe crowding (LII ≥ 3 mm), with no labio-lingually displaced teeth
* Class I or Class II malocclusion by ½ cusp or less
* Non-extraction in both arches
* Age 11-60
* Good oral hygiene
* Non-smoker; non-use of chewing tobacco

Exclusion Criteria:

* Subject is currently enrolled in another clinical study
* Subject decided on Invisalign rather than braces
* Periodontally involved teeth
* Use of bisphosphonates (osteoporosis drugs) during the study
* Subject plans to relocate over the treatment period
* Spaces between anterior teeth
* Subject has dental implants or an implanted prosthesis
* Sponsor employees, the Investigator and staff, as well as their immediate family members

Ages: 11 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Rate of tooth movement in OrthoPulse treated and non-OrthoPulse treated patients | From start of treatment until Little's Irregularity Index (LII) reaches less than approximately 2 mm but greater than 0 mm, no more than 6 months after the start of treatment.
  Rate of tooth movement will be evaluated based on the duration of time and amount of tooth movement required to reach Little's Irregularity Index (LII) of less than approximately 2 mm but greater than 0 mm, as determined by the qualified investigator.

SECONDARY OUTCOMES:
Effect of OrthoPulse PBM on external apical root resorption (EARR) | 6 months after the start of orthodontic treatment
  Root lengths from patients will be measured using panoramic radiographs at the start of treatment and 6 months after the start of treatment. These measurements will be used to determine and compare EARR between each of the two groups.
Risk of OrthoPulse PBM to the patient. | Participants will be followed for the duration of their orthodontic treatment, an expected average of 1-2 years, depending on the severity of the case
  Patients from both groups will be questioned and assessed at regularly scheduled visits for treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brawn, DDS, Study Director — Biolux Research Holdings, Inc.
Locations (3):
- United States (3):
  - Dickerson Orthodontics, Chandler, Arizona
  - Dickerson Orthodontics, Peoria, Arizona
  - Dickerson Orthodontics, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Background] Sun X, Zhu X, Xu C, Ye N, Zhu H. [Effects of low energy laser on tooth movement and remodeling of alveolar bone in rabbits]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2001 Oct;19(5):290-3. Chinese. PMID 12539482
- [Background] Yamaguchi M, Hayashi M, Fujita S, Yoshida T, Utsunomiya T, Yamamoto H, Kasai K. Low-energy laser irradiation facilitates the velocity of tooth movement and the expressions of matrix metalloproteinase-9, cathepsin K, and alpha(v) beta(3) integrin in rats. Eur J Orthod. 2010 Apr;32(2):131-9. doi: 10.1093/ejo/cjp078. Epub 2010 Feb 16. PMID 20159792
- [Background] Nimeri G, Kau CH, Corona R, Shelly J. The effect of photobiomodulation on root resorption during orthodontic treatment. Clin Cosmet Investig Dent. 2014 Jan 15;6:1-8. doi: 10.2147/CCIDE.S49489. eCollection 2014. PMID 24470774
- [Background] Ekizer A, Uysal T, Guray E, Akkus D. Effect of LED-mediated-photobiomodulation therapy on orthodontic tooth movement and root resorption in rats. Lasers Med Sci. 2015 Feb;30(2):779-85. doi: 10.1007/s10103-013-1405-3. Epub 2013 Aug 29. PMID 23990217
- [Background] Ekizer A, Uysal T, Guray E, Yuksel Y. Light-emitting diode photobiomodulation: effect on bone formation in orthopedically expanded suture in rats--early bone changes. Lasers Med Sci. 2013 Sep;28(5):1263-70. doi: 10.1007/s10103-012-1214-0. Epub 2012 Nov 9. PMID 23139069
- [Background] El-Bialy T, Alhadlaq A, Felemban N, Yeung J, Ebrahim A, Hassan AH. The effect of light-emitting diode and laser on mandibular growth in rats. Angle Orthod. 2015 Mar;85(2):233-8. doi: 10.2319/030914-170.1. Epub 2014 Jul 14. PMID 25017014
- [Background] Uysal T, Ekizer A, Akcay H, Etoz O, Guray E. Resonance frequency analysis of orthodontic miniscrews subjected to light-emitting diode photobiomodulation therapy. Eur J Orthod. 2012 Feb;34(1):44-51. doi: 10.1093/ejo/cjq166. Epub 2010 Dec 27. PMID 21187526
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Shaughnessy T, Kantarci A, Kau CH, Skrenes D, Skrenes S, Ma D. Intraoral photobiomodulation-induced orthodontic tooth alignment: a preliminary study. BMC Oral Health. 2016 Jan 13;16:3. doi: 10.1186/s12903-015-0159-7. PMID 26762247
- [Background] Doshi-Mehta G, Bhad-Patil WA. Efficacy of low-intensity laser therapy in reducing treatment time and orthodontic pain: a clinical investigation. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):289-297. doi: 10.1016/j.ajodo.2011.09.009. PMID 22381489
- [Background] Dias FJ, Issa JP, Vicentini FT, Fonseca MJ, Leao JC, Siessere S, Regalo SC, Iyomasa MM. Effects of low-level laser therapy on the oxidative metabolism and matrix proteins in the rat masseter muscle. Photomed Laser Surg. 2011 Oct;29(10):677-84. doi: 10.1089/pho.2010.2879. Epub 2011 Jul 11. PMID 21745137
- [Background] Silveira PC, Silva LA, Fraga DB, Freitas TP, Streck EL, Pinho R. Evaluation of mitochondrial respiratory chain activity in muscle healing by low-level laser therapy. J Photochem Photobiol B. 2009 May 4;95(2):89-92. doi: 10.1016/j.jphotobiol.2009.01.004. Epub 2009 Jan 21. PMID 19232497
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Sousa MV, Scanavini MA, Sannomiya EK, Velasco LG, Angelieri F. Influence of low-level laser on the speed of orthodontic movement. Photomed Laser Surg. 2011 Mar;29(3):191-6. doi: 10.1089/pho.2009.2652. Epub 2011 Jan 23. PMID 21254890
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Weber JB, Pinheiro AL, de Oliveira MG, Oliveira FA, Ramalho LM. Laser therapy improves healing of bone defects submitted to autologous bone graft. Photomed Laser Surg. 2006 Feb;24(1):38-44. doi: 10.1089/pho.2006.24.38. PMID 16503787
- [Background] Oron U, Ilic S, De Taboada L, Streeter J. Ga-As (808 nm) laser irradiation enhances ATP production in human neuronal cells in culture. Photomed Laser Surg. 2007 Jun;25(3):180-2. doi: 10.1089/pho.2007.2064. PMID 17603858
- [Background] Masha RT, Houreld NN, Abrahamse H. Low-intensity laser irradiation at 660 nm stimulates transcription of genes involved in the electron transport chain. Photomed Laser Surg. 2013 Feb;31(2):47-53. doi: 10.1089/pho.2012.3369. Epub 2012 Dec 16. PMID 23240874